CLINICAL TRIAL: NCT03288168
Title: Multi-center Retrospective Study on Clinical Features and Molecular Subgroups of Children and Adolescents With Medulloblastoma in China
Brief Title: Children's and Adolescents' Medulloblastoma Molecular Subgroups in China
Acronym: CNOG-MB001
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Children's Neuro-Oncology Group (CNOG) (Unknown)
Responsible Party: Principal Investigator, Jie Ma, MD, PhD, Head of Department of Pediatric Neurosurgery, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-17-014; CNOG-MB001 (Other: Children's Neuro-Oncology Group)
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Medulloblastoma, Childhood
Keywords: Observation; Molecular Subgroup; NanoString
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Either paraffin embedded tissue block or frozen tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 0-18 y/o Patients with Medulloblastoma: Patients treated with comprehensive treatments including surgery, chemo-therapy with / without (less than 3 y/o) radiation, during the period of Jan 2008 and Dec 2012, whose tumor samples will be tested by NanoString and Histochemistry methods, are enrolled in this cohort group.

SUMMARY:
Recently, diagnosis and treatments for medulloblastoma becomes more complicated than before since the new World Health Organization (WHO) diagnosis criteria has put molecular marker onto an ever important position. Reports and studies revealed highly correlated connection between subgroups of medulloblastoma and patient outcomes. Children's Oncology Group (COG) has launched many new studies on molecular subgroups-based specific treatment trails. In China, children and adolescents with brain tumor have been treated variously for a long time in lack of standardized comprehensive treatments. Same poor situation in basic research and clinical studies makes the Chinese children with brain tumor hardly catch up with international level in molecular diagnosis and specific treatments. There are limited studies, which were conducted by immunohistochemistry for identifying medulloblastoma molecular subgroups, indicating the similar correlation of the subgroups and outcomes to world-wide reports. As the Children's Neuro-Oncology Group (CNOG) was established in China in May 2017, it makes studies from multiple centers in children's brain tumors become practical. And the availability of DNA methylation array, NanoString and other methods in medulloblastoma subgroup identification assures the quality of the method for this study.

DETAILED DESCRIPTION:
Studies discovered that medulloblastoma is a group of tumors with different pathogenesis through different pathways, and majorly can be divided into four molecular subgroups. Moreover, multicenter retrospective studies from US, Canada and European Countries revealed that the molecular subgroup of medulloblastoma becomes an independent correlated risk factor for the patient outcomes. This finding made WHO classification of tumours of central nervous system consider the markers in molecular pathway be an ever important indicator in the new diagnosis criteria. In COG prospective studies for target therapies, subgroup distinguishing becomes indispensable, and the use of immunohistochemistry combined with NanoString, DNA methylation arrays or other molecular methods makes subgroup identification more reliable. In China, there are limited single institutional studies, which were all conducted by immunohistochemistry or polymerase chain reaction (PCR), on molecular sub-grouping of medulloblastoma, especially in pediatric patients. This multicenter retrospective study enrolls children and adolescents (0-18y/o) with primary medulloblastoma from CNOG member institutions across the country, with available paraffin embedded samples and reliable follow-up information, to assess the correlation of molecular subgroups of medulloblastoma and outcomes in Chinese population.

This multicenter study recruits eligible patients from CNOG member institutions. Data validation and verification is double conducted by each center and investigators in central data base. Case report form (CRF) was designed by principle investigator and will be modified in the period of uploading first 5 cases by each participated center. The estimated enrollment is 200 cases after sample size assessment. Descriptive statistical analysis, Two-Sample (Independent group) T-Test and one-way ANOVA will be used in epidemiological analysis. Cox-regression / Kaplan-Meier plot will be used in survival analysis. Chi-square test will be used to validate the test efficiency of immunohistochemistry and NanoString methods.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have classical histology posterior fossa medulloblastoma as determined by institutional neuro-pathological evaluation.
* Participants must have tumor tissue samples (either paraffin embedded tissue block or frozen tissue) for NanoString test for distinguishing the molecular subgroups of medulloblastoma in Xinhua hospital affiliated to Shanghai Jiaotong University School of Medicine (SHXH).
* Participants must provide tumor tissue samples (either paraffin embedded tissue block or frozen tissue) for immunohistochemistry assessment in verifying the molecular subgroups of medulloblastoma, or conduct the same immunohistochemistry test according to central analysis in SHXH, and send the slides to SHXH for center reviewing.
* Diagnostic imaging (pre and post operation (OP) contrast MRI or CT, Post-OP imaging conducted within 72 hours, no later than 14 days) must be forwarded to SHXH for central review to confirm eligibility.
* Sufficient pathologic material must be available for central analysis and review in SHXH.
* The patients must have no previous radiotherapy or chemotherapy other than corticosteroids.
* Ability to understand and willingness to comply with follow-up visits.
* Life expectancy more than 4 weeks.

Exclusion Criteria:

* Patients must not have received any prior tumor-directed therapy other than surgical intervention and corticosteroids.
* Tumor tissue sample not available for biological studies (from the initial diagnosis and/or relapse).
* Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate standard treatment or would likely interfere with study results.
* Patients obtained no radiation and/or chemo therapies are not excluded in this study since the nature history of the disease will also be evaluated.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents from 0-18 y/o, diagnosed with Medulloblastoma in CNOG-MB001 study participated institutions in mainland China, with available detailed clinical records, full followup records and available tumor samples, fitting eligibility criteria, are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Follow-up for final survival period till 31 December 2017 or last available contact, whichever occurred first
  The observation period of outcome started with the first medical record available on site till last contact available on site or the end of the observation period (31 December 2017), whichever occurred first.

SECONDARY OUTCOMES:
Event Free Survival | Follow-up for none-recurrence survival (metastasis/relapse) period till 31 December 2017 or last available contact, whichever occurred first.
  The observation period of outcome started with the first medical record available on site till last contact available on site or the end of the observation period (31 December 2017), whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jie MA, MD, Phd, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (9):
- China (9):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fuzhou General Hospital of Nanjing Military Region, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong 999 Brain Hospital, Guangzhou, Guangdong
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided